CLINICAL TRIAL: NCT03176433
Title: A Multicentre, Single-arm, Prospective Clinical Trial to Investigate the Safety and Feasibility of Cold Storage Prior to Normothermic Machine Perfusion in Adult Human Liver Transplantation
Brief Title: Post Static Cold Storage Normothermic Machine Liver Perfusion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/LO/2196
Record Dates: First submitted 2017-05-04; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Normothermic Machine Liver Perfusion — Liver Preservation Method

SUMMARY:
The aim of this study is to assess the safety and feasibility of a short period of cold storage prior to normothermic machine perfusion in adult liver transplantation.

ELIGIBILITY:
Donor Inclusion Criteria:

* Donors over the age of 16 years.
* Liver allografts from donation after brain death (DBD), standard and extended criteria donors. (SCD, ECD) and donation after circulatory death (DCD) donors.
* Liver must be perfused on OrganOx metra perfusion device within 8 hours of in situ cold perfusion.
* The perfusion should last a minimum of 4 hours and maximum of 24 hours.

Donor Exclusion Criteria:

* Living donors.
* Liver being transplanted as part of a multi-organ transplant (eg liver and kidney).
* Liver intended for split transplant.
* Donor age <16 years
* Liver which investigator is unwilling to recruit to study.
* Any liver in which logistics prevent perfusion on the OrganOx metra perfusion device within 8 hours of in situ cold perfusion.

Recipient Inclusion Criteria:

* Adult patients (18 years or more).
* Active on the waiting list for liver transplantation.
* Able to give informed consent.

Recipient Exclusion Criteria:

* Age less than 18 years.
* Acute/fulminant liver failure.
* Transplantation of more than one organ (e.g. liver and kidney).
* Refusal of informed consent.
* Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient and Graft Survival | 30 days
  Patient survival after liver transplantation and liver graft survival will be assessed at 30-days post-op as a composite outcome measure. This will be recorded as yes/no outcome.

SECONDARY OUTCOMES:
Peak serum AST (U/L) | 7 days
  The highest AST level recorded in the first 7 days post-transplant will be identified. This is a surrogate marker for longer-term outcome. It will be compared with matched controls of livers undergoing continuous NMP and SCS
Early allograft dysfunction (EAD) | 7 days
  This is a composite score which is used to predict longer-term outcome. It comprises: bilirubin >or=10mg/dL on day 7 post-transplant, international normalized ratio >or=1.6 on day 7 post-transplant, and alanine or aspartate aminotransferases >2000 IU/L within the first 7 days post-transplant. This will be compared with matched controls of livers undergoing continuous NMP and SCS
Primary non-function | 10 days
  This is irreversible graft dysfunction requiring emergency liver replacement during the first 10 days after liver transplantation, in the absence of technical or immunological causes.
  This will be compared with matched controls of livers undergoing continuous NMP and SCS
Adverse events, transplantation and organ discard rates. | 30 days
  This composite outcome aims to establish safety and feasibility as well as organ utilisation. It will be compared with matched controls of livers undergoing continuous NMP and SCS
Biliary investigation or intervention | 6 months
  In order to capture the incidence of ischaemic cholangiopathy, any biliary investigation (such as magnetic resonance imaging) or intervention (such as endoscopic retrograde cholangiopancreatography) will be recorded and compared with matched controls of livers undergoing continuous NMP and SCS
Patient and Graft Survival | 6 months
  Patient survival after liver transplantation and liver graft survival will be assessed at 6 months post-op as a composite outcome measure. This will be recorded as yes/no outcome and compared controls undergoing continuous NMP and SCS
Patient and Graft Survival | 12 months
  Patient survival after liver transplantation and liver graft survival will be assessed at 12 months post-op as a composite outcome measure. This will be recorded as yes/no outcome and compared controls undergoing continuous NMP and SCS

CONTACTS AND LOCATIONS:
Overall Officials: Peter Friend, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - King's College Hospital, London
  - Royal Free Hospital, London